CLINICAL TRIAL: NCT05854784
Title: Proof of Concept, Phase IIa, Open Label Study to Evaluate the Safety and Efficacy of Afamelanotide in Patients With Variegate Porphyria (VP)-Related Skin Disease.
Brief Title: Study to Evaluate the Safety and Efficacy of Afamelanotide in Patients With Variegate Porphyria (VP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUV040
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Variegate Porphyria
MeSH Terms: conditions — Porphyria, Variegate | interventions — afamelanotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Afamelanotide (Experimental)
  Interventions: Drug: Afamelanotide 16 MG

INTERVENTIONS:
Drug: Afamelanotide 16 MG — Eligible patients will receive one dose of afamelanotide 16mg every 28 days (up to six doses), as a controlled-release formulation.

SUMMARY:
The primary objective is to evaluate the impact of afamelanotide on the severity of skin disease in patients with Variegate Porphyria (VP). The secondary objectives are to evaluate the safety and tolerability of afamelanotide in patients with VP and evaluate the impact of afamelanotide on the quality of life of patients with VP.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with confirmed diagnosis of VP.
* Patients with VP-related skin symptoms.
* Aged 18-70 years.

Exclusion Criteria:

* Allergy to afamelanotide or polymer or to local anaesthetic to be used if applicable.
* Had two or more acute attacks of hepatic porphyria, as defined by the occurrence or acute porphyric symptoms within 12 months prior to the Screening period.
* Individual history of malignant or premalignant skin lesions.
* Individual or family history of melanoma.
* Presence of severe hepatic disease.
* Renal impairment.
* Female who is pregnant or lactating.
* Females of child-bearing potential not using adequate contraceptive or a life-style excluding pregnancy.
* Sexually active man with a partner of child-bearing potential not using adequate contraceptive measures.
* Use of any other prior and concomitant therapy which may interfere with the objective of the study, within 30 days prior to the Screening period.
* Participation in a clinical trial within 30 days prior to the Screening period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CLINUVEL investigational site, Rotterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- SCENESSE® (Afamelanotide 16mg): Six eligible patients received one dose of afamelanotide 16mg every 28 days, 6 doses in total, as a controlled-release formulation.
Period: Overall Study
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1
  Race: White (non-Hispanic, Latino or Spanish) | 4
  Race: White (Hispanic, Latino or Spanish) | 1
Confirmed diagnosis of Varigate Porphyria [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: The Change in Disease Severity in Patients With VP as Measured by CGIC.
Description: The higher the score, the less severe the disease. Scale ranges from +3 to -3.
Time Frame: From baseline to Day 168
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Afamelanotide
Number analyzed (Participants) | 6
Scores on a scale | 2.5 [1.0 to 3.0]

2. Secondary Outcome: The Change in Disease Severity in Patients With VP as Measured by 11-point VAS IGA.
Description: A lower score indicates a reduced severity of the disease.Scale ranges from 0 to 10.
Time Frame: Median change from baseline to Day 168.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Scores on a scale | -3.0 [-5.0 to 0.0]

3. Secondary Outcome: The Change in Disease Severity in Patients With VP as Measured by 5-point IGA.
Description: A lower score indicates a reduced severity of the disease. Scale ranges from 0 to 4.
Time Frame: Median change from baseline to Day 168
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Scores on a scale | -2.0 [-3.0 to 1.0]

4. Secondary Outcome: The Change in Disease Severity in Patients With VP as Measured by PGIC.
Description: The higher the score, the less severe the disease. Score ranges from +3 to -3.
Time Frame: Median change from baseline to Day 168
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Scores on a scale | 2.5 [1.0 to 3.0]

5. Secondary Outcome: The Change in Disease Severity in Patients With VP as Measured by PGA Using VAS.
Description: A lower score indicates a reduced severity of the disease. Scale ranges from 0 to 10.
Time Frame: Median change from baseline to Day 168
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Scores on a scale | -6.5 [-9.0 to -1.0]

6. Secondary Outcome: The Change in Number of New Skin Lesions Formed.
Description: A lower number indicates a reduced severity of the disease.
Time Frame: Median change from baseline to Day 168.
Measure: Median (Full Range); unit: Lesions
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Lesions | -6.5 [-11.0 to 4.0]

7. Secondary Outcome: The Change in the Quality of Life in Patients With VP as Measured by WPAI:GH.
Description: Higher score indicates greater impairment and less productivity. Score is percentage impairment.
Time Frame: Median of change from baseline to Day 168
Measure: Median (Full Range); unit: Percentage of impairment time
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Percentage of impairment time | -10.00 [-80.0 to 40.0]

8. Secondary Outcome: The Change in the Quality of Life in Patients With VP as Measured by VP-derived QOLEB.
Description: Higher scores represent worse health-related quality of life. Scale ranges from 0 to 45.
Time Frame: From baseline to Day 168
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Score on a scale | -12.0 [-23.0 to -3.0]

9. Secondary Outcome: The Change in the Quality of Life in Patients With VP as Measured by VP QoL.
Description: "Quality of life measured by the number of responses of "much better than a year ago" to the question "How would you judge the condition of your skin of your face and hands today, in comparison to the situation last year (12 months ago)?"
Time Frame: Assessed at baseline and Day 168 to reflect retrospective changes over the previous 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Participants
  Baseline | 0
  Day 168 | 5

10. Secondary Outcome: The Change in Outdoor Light Exposure Over Time (Daily Diary)
Description: Daily diaries recording outdoor light exposure.
Time Frame: From baseline to Day 168.
Measure: Median (Full Range); unit: Change in number of hours of sunlight
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Change in number of hours of sunlight | 0.70 [0.2 to 2.3]

ADVERSE EVENTS:
Time Frame: All adverse events were monitored from baseline until 3 months after end of treatment (approximately 9 months)
Description: AE are reported as "General Disorders" to maintain confidentiality as the patients in this study are European Union citizens.The European Medicines Agency (EMA) has agreed that where single patient adverse event cases occur in a rare disease study there is a potential for identification of the patient.The EMA therefore considers such AE cases to be medical information on an individual and accepts redaction of the information on General Data Protection Regulation (Regulation(EU)2016/679) grounds.
Arm/Group | SCENESSE® (Afamelanotide 16mg)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCENESSE® (Afamelanotide 16mg) (N=6)
General disorders (General disorders) | 4 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT05854784/Prot_SAP_001.pdf